CLINICAL TRIAL: NCT06262945
Title: Comparative Examination of the Postoperative Effects of Low-laser Treatment and Platelet-rich Fibrin Applications After Mandibular Impacted Wisdom Teeth Extraction
Brief Title: Comperasion the Postoperative Effect of Low Laser Therapy and Platelet Rich Fibrin on Mandibular Third Molar Surgery.
Status: Completed | Type: Observational
Sponsor: Beste Erismen (Other)
Responsible Party: Sponsor-Investigator, Beste Erismen, Phd Stıdent, Near East University, Turkey
Organization: Near East University, Turkey (Other)
Other Study IDs: YDU/2024/120-1808
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Impacted Third Molar Tooth
Keywords: platelet rich fibrin; comparison; low laser therapy; wisdom tooth
MeSH Terms: interventions — Diagnosis; Penicillins; Analgesics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: platelet rich fibrin placed into the socket of the extraciton tooth + Augmentin 1gr tablet prescribed 2 times a day
  Interventions: Diagnostic Test: Diagnoses; Procedure: traditional osteotomies; Biological: platelet rich fibrin; Drug: Antibiotics, Penicillin; Drug: Analgesic
- Group 2: platelet rich fibrin placed in to the socket of the extractraciton tooth combined with low laser treatment extraorally to the extraction area for three days within surgery day + Augmentin 1gr tablet prescribed 2 times a day
  Interventions: Diagnostic Test: Diagnoses; Procedure: traditional osteotomies; Biological: platelet rich fibrin; Drug: Antibiotics, Penicillin; Device: low laser therapy, bicure laser; Drug: Analgesic
- Group 3: Low Laser Treatment was applied to the extraorally to the extraction area for three days within surgery day + Augmentin 1gr tablet prescribed 2 times a day
  Interventions: Diagnostic Test: Diagnoses; Procedure: traditional osteotomies; Drug: Antibiotics, Penicillin; Device: low laser therapy, bicure laser; Drug: Analgesic
- Control group.: Tradional osteomy was made. + Augmentin 1gr tablet prescribed 2 times a day
  Interventions: Diagnostic Test: Diagnoses; Procedure: traditional osteotomies; Drug: Antibiotics, Penicillin; Drug: Analgesic

INTERVENTIONS:
Diagnostic Test: Diagnoses — All of the patients withstand a radiological examination, including panoramic radiography, and all were handled by the same surgeon and assistant.
Procedure: traditional osteotomies — In all groups the flap incision was triangular in shape which avoids muscle involvement (Archer flap).
Biological: platelet rich fibrin — Platelet rich fibrin (PRF), is an example and popular procedure for accelerate healing of soft and hard tissue because of the presence of various growth factors.a blood sample was taken without anticoagulant in 10 mL glass-coated plastic tubes that were immediately centrifuged (Elektro-mag M415P) at 3,000 rpm for 10 min (approximately 400 g) (13). The platelet-poor plasma that accumulated at the top of the tubes was discarded.PRF was dissected approximately 2 mm below its contact point with the red corpuscles situated beneath, to include any remaining platelets that may have localized below the junction between the PRF and red corpuscles.
  Groups: Group 1; Group 2
Drug: Antibiotics, Penicillin — Antibiotics are prescribed for the patients.
Device: low laser therapy, bicure laser — There are studies in the literature that low-energy lasers have positive effects on the biological and biochemical processes of wound healing. Acceleration of local circulation, increase in cell proliferation and collagen synthesis are among the various effects of laser application. B Cure Dental Pro Laser application will be applied to the patient for the first 3 days. Low dose laser application will be applied to the angulus area, covering the surgical area for 8 minutes. Before this laser procedure, the patient will be asked to fill out a pain scale. This pain scale and the number of analgesics used will be monitored for 3 days.
  Groups: Group 2; Group 3
Drug: Analgesic — Analgesics are prescribed for the patients.

SUMMARY:
The aim of this study was investigate the comparison of postoperative effects of low laser treatment and platelet-rich fibrin application on mandibular impacted third molar tooth extraction. The study included a total of 60 patients with impacted mandibular third molar. Patients were evaluated in 4 randomly separated groups. In group 1, PRF was applied to the tooth socket. In group 2, PRF was applied to the tooth socket combined with Low Laser Treatment extraorally to the extraction area for three days within surgery day In group 3, Low Laser Treatment was applied to the extraorally to the extraction area for three days within surgery day. In group 4 (control group), tradional osteomy was made. The outcome variables were pain, swelling, the number of analgesics taken, and trismus. These variables were also assessed based on first, second, third, and seventh days following the operation. All of the 4 groups patients were prescribed an 875/125 mg amoxicillin/clavulanic acid tablet twice daily for five days.

ELIGIBILITY:
Inclusion Criteria:

* The patient had no systemic diseases, no taken opioids for a long period, no current infections or acute pericoronitis, no smoke or drink alcohol, no pregnancy, the absence of allergy to penicillin and presence of penicillin allergy.

Exclusion Criteria:

* pericoronitis, no inflammation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community aged between 18-40 without any important systemic disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | Day 1
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
Visual analogue scale (VAS) | Day 2
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
Visual analogue scale (VAS) | Day 3
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
Visual analogue scale (VAS) | Day 7
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
Trismus | Day 1
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
Trismus | Day 2
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
Trismus | Day 3
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
Trismus | Day 7
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
Swelling | Day 1
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.
Swelling | Day 2
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.
Swelling | Day 3
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.
Swelling | Day 7
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.

SECONDARY OUTCOMES:
the number of analgesic tablets | Day 1
the number of analgesic tablets | Day 2
the number of analgesic tablets | Day 3
the number of analgesic tablets | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Beste Erismen Agan, Principal Investigator — Near East University
Locations (1):
- Near East University, Nicosia, Lefkosa, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desmet KD, Paz DA, Corry JJ, Eells JT, Wong-Riley MT, Henry MM, Buchmann EV, Connelly MP, Dovi JV, Liang HL, Henshel DS, Yeager RL, Millsap DS, Lim J, Gould LJ, Das R, Jett M, Hodgson BD, Margolis D, Whelan HT. Clinical and experimental applications of NIR-LED photobiomodulation. Photomed Laser Surg. 2006 Apr;24(2):121-8. doi: 10.1089/pho.2006.24.121. PMID 16706690
- [Background] Krynicka I, Rutowski R, Staniszewska-Kus J, Fugiel J, Zaleski A. The role of laser biostimulation in early post-surgery rehabilitation and its effect on wound healing. Ortop Traumatol Rehabil. 2010 Jan-Feb;12(1):67-79. PMID 20203347
- [Background] Donmezer CM, Bilginaylar K. Comparison of the Postoperative Effects of Local Antibiotic versus Systemic Antibiotic with the Use of Platelet-Rich Fibrin on Impacted Mandibular Third Molar Surgery: A Randomized Split-Mouth Study. Biomed Res Int. 2021 Dec 2;2021:3040661. doi: 10.1155/2021/3040661. eCollection 2021. PMID 34901267
- [Background] Feslihan E, Eroglu CN. Can Photobiomodulation Therapy Be an Alternative to Methylprednisolone in Reducing Pain, Swelling, and Trismus After Removal of Impacted Third Molars? Photobiomodul Photomed Laser Surg. 2019 Nov;37(11):700-705. doi: 10.1089/photob.2019.4696. Epub 2019 Oct 7. PMID 31589558
- [Derived] Erismen Agan B, Uyanik LO, Donmezer CM. Comparison of the postoperative effect of low laser therapy and platelet rich fibrin on mandibular third molar surgery: a randomized study. BMC Oral Health. 2025 Mar 25;25(1):427. doi: 10.1186/s12903-025-05828-3. PMID 40134000